CLINICAL TRIAL: NCT02968485
Title: A Phase I, Open Label, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SHR7390 in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of SHR7390 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR7390-I-101-AST
Record Dates: First submitted 2016-10-07; First posted 2016-11-18 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumor
Keywords: advanced solid tumor; Protein Kinase MEK inhibitor (MEKi); Safety; Pharmacokinetics
MeSH Terms: interventions — MEK inhibitor I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHR7390 (Experimental): 60 subjects with advanced solid tumors were received single and then multiple oral doses of SHR7390(2 cycles,each cycle 28days).
  Interventions: Drug: SHR7390

INTERVENTIONS:
Drug: SHR7390 — SHR7390 is provided as white, film-coated,immediate release tablets containing SHR7390 at dosage strengths of 0.125 mg and 0.5 mg. Multiple tablets of SHR7390 will be administered daily to achieve targeted doses of SHR7390: 0.25 mg-4 mg. Tablets will be orally administered with 240 ml water, once daily, 2 hours after a meal.
  Other Names: MEK inhibitor

SUMMARY:
This aim of study to assess the safety and tolerability of SHR7390 and to define the maximum tolerated dose (MTD) of SHR7390 in the patients with advanced solid tumors.

To evaluate the pharmacokinetics of SHR7390 in patients with advanced solid tumors.

To study the effects of food on the pharmacokinetic parameters of SHR7390. To assess the antitumor activity of SHR7390 in patients with advanced solid tumors preliminarily and recommend reasonable dosage regimen for the follow-up clinical trial.

DETAILED DESCRIPTION:
This is an open-label, dose escalation study of repeated doses of SHR7390 in the patients with advanced solid tumors that have no targeted agent as standard of therapy.

A study cycle is defined as SHR7390 administered once daily orally for 28 days. Dose limiting toxicities (DLT) will be assessed in the first cycle of treatment. the trial is dose escalation and is designed by Accelerated Titration Designs during initial accelerated phase. when the significant toxicity or DLT is observed in any course of treatment,the accelerated titration trial terminates and subsequent cohort sizes and dose escalation are a conventional design of 3+3 patients. If one adverse event （AE） meets dose limiting toxicity (DLT) criteria at a given dose, 3 additional patients will be enrolled in this dose cohort. If 2 DLTs are determined at a given dose level, this dose will be designated as the MTD.

Additional patients will be enrolled for PK evaluations at different dose levels based on preliminary safety and tolerability. Multiple blood samples at designated time points will be collected for PK evaluations.

The safety, tolerability and AEs will be closely monitored throughout the study duration. The preliminary effectiveness and clinical benefits of SHR7390 will be evaluated as a single agent.

The evaluation of the effects of a high-fat, high-calorie meal on the single-dose pharmacokinetics (PK) of SHR7390.The design to assess food-effect is a randomized, balanced, 2-treatment(fed vs. fasted), separated by an adequate wash-out period.

ELIGIBILITY:
Inclusion Criteria:

The study is open to all males and females who meet the following inclusion criteria at screening and baseline to participate in the study.

To be included to participate in this study each patient must:

1. 18-70 years of age, both women and men;
2. invalid the standard treatment or non standard and effective treatment in patients with advanced solid tumors diagnosed by pathology;
3. the Eastern Cooperative Oncology Group （ECOG） General status (performance status, PS) of 0-1;
4. the expected lifetime ≥ 3 months;
5. organ function you must meet the following requirements:

   * Adequate bone marrow reserve: including neutrophil absolute count,platelets and hemoglobin;
   * Liver: serum albumin ≥ 3.0 g/dl; bilirubin, Alanine aminotransferase（ALT）and aspartate aminotransferase（AST）≤ 1.5 x upper limit of normal value (ULN),if there is liver metastasis, the ALT or AST

     * 5x upper limit of normal value (ULN);
   * Kidneys: creatinine clearance ≥ 50 mL/min (Cockcroft-Gault of the standard formula）；
   * Heart: left ventricular ejection fraction ≥ 50%; normal Electrocardiograph (ECG) and corrected QT interval（QTc）;
6. The damage of the patients caused by other treatments has been restored;
7. A agreement to use a highly effective, non-hormonal form of contraception is required for women of childbearing potential and men with partners of childbearing potential, who were not sterilized surgically, for duration of the study treatment and after the last dose of study treatment; For female patients of child bearing potential,who was not sterilized surgically,the serum human chorionic gonadotropin （HCG） pregnancy test must be the negative
8. Written informed consent is provided by signing the informed consent form.

Exclusion Criteria:

Subjects who meet any of the criteria listed below will not be eligible for participation in this study. A patient will not be eligible for study participation if:

1. Previous treatment with other protein kinase MEK inhibitors;
2. Use of other investigational anti-cancer drugs or the termination of the investigational drugs within the last four weeks;
3. Currently or possibly receiving other cancer therapy during the study period;
4. Presence of a factor that influences the oral drug (such as inability to swallow) or presence of active gastrointestinal disease or other conditions that will interfere significantly with the absorption, distribution, metabolism, or excretion of drug;
5. History of retinal vascular occlusion （RVO） or central serous retinopathy;
6. Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for retinal vein thrombosis or central serous retinopathy;
7. Intraocular pressure>21mmHg as measured by tonography or glaucoma;
8. Tumor metastases of central nervous system or leptomeningeal metastases. primary malignancy of the central nervous system;
9. Evidence of severe or uncontrolled systemic diseases (e.g. unstable or uncompensated respiratory, hepatic, renal or cardiac diseases);
10. History of acute coronary syndromes (including unstable angina);
11. Presence of arrhythmia, myocardial ischemia with drug intervention. III-IV stage heart failure as defined by the New York Heart Association (NYHA) functional classification system.
12. Medical treatment for an acute phase of infection;
13. hepatitis B virus（HBV) or hepatitis C virus (HCV) infection stage with abnormal liver function;
14. History of immunodeficiency, or other acquired and congenital immunodeficiency disease;
15. Psychological, familial, sociological or geographical conditions that do not permit compliance with protocol;
16. Unwillingness or inability to follow the procedures outlined in the protocol;
17. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Day 1 to 28 ( Cycle 1)
  to assess safety and tolerability of SHR7390 with a maximum tolerated dose (MTD) of SHR7390 in patients with advanced solid tumors

SECONDARY OUTCOMES:
The measurement of maximum plasma concentration (Cmax) | Up to 2 cycles(each cycle 28 days)
The measurement of the area under the plasma concentration-time versus time curve(AUC) | Up to 2 cycles(each cycle 28 days)
The measurement of elimination half life (T1/2) | Up to 2 cycles(each cycle 28 days)
The measurement of time of maximum plasma concentration (Tmax) | Up to 2 cycles(each cycle 28 days)
The Measurement of mean retention time (MRT) | Up to 2 cycles(each cycle 28 days)
The measurement of apparent volume of distribution (Vd) | Up to 2 cycles(each cycle 28 days)
The measurement of clearance (Cl) | Up to 2 cycles(each cycle 28 days)
The measurement of linear Relationship | Up to 2 cycles(each cycle 28 days)
The measurement of drug accumulation ratio | Up to 2 cycles(each cycle 28 days)
The comparison of maximum plasma concentration (Cmax) in the fed and fasted states | 2 weeks
The comparison of the area under the plasma concentration-time versus time curve(AUC) in the fed and fasted states | 2 weeks
The comparison of elimination half life(T1/2) in the fed and fasted states | 2 weeks
The comparison of time of maximum concentration (Tmax) in the fed and fasted states | 2 weeks
The comparison of mean retention time (MRT) in the fed and fasted states | 2 weeks
The comparison of apparent volume of distribution (Vd）in the fed and fasted states | 2 weeks
The comparison of clearance (Cl) in the fed and fasted states | 2 weeks
The comparison of AUC 0-24h in the fed and fasted states | 2 weeks
The imaging data of the subjects will be evaluated at the ends of cycle 1 and cycle 2 by RECIST1.1 evaluation criteria separately. | 2 cycles(each cycle 28 days)
Response rate objective (ORR) will be evaluated at the different dose levels | 2 cycles(each cycle 28 days)
Disease control rate (DCR) will be evaluated at the different dose levels | 2 cycles(each cycle 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: RuiHua Xu, MD, PhD, Principal Investigator — The Cancer Center,Sun Yat-sen University
Locations (1):
- The Cancer Center,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No